CLINICAL TRIAL: NCT01071447
Title: Nurse-led Clinic for Patients With Rheumatic Diseases and Biological Treatment:a Randomized Controlled Trial Comparing Nurse-led Clinic Versus Rheumatologist Clinic
Brief Title: Nurse-led Clinic for Patients With Rheumatic Diseases and Biological Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spenshult Hospital (Other)
Collaborators: The Swedish Rheumatism Ass (Other); County Council of Halland, Sweden (Other Government)
Responsible Party: Stefan Bergman, Research Director, R&D-centre Spenshult Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FoUS09001
Record Dates: First submitted 2009-10-08; First posted 2010-02-19 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Rheumatic Diseases
Keywords: Rheumatic diseases; Biologic treatment; Nurse-led
MeSH Terms: conditions — Rheumatic Diseases | interventions — Practice Patterns, Nurses'

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rheumatologist-led clinic (Active Comparator): Rheumatologist-led clinic: The subjects are seeing a rheumatologist after six months and after 12-months of intervention and have the possibility to contact the rheumatology clinic
  Interventions: Other: Nurse-led clinic vs rheumatologist-led clinic
- Nurse-led clinic (Experimental): The subjects are seeing a rheumatology nurse after six months and a rheumatologist after 12 months of intervention and have the possibility to contact the rheumatology nurse during the intervention.
  Interventions: Other: Nurse-led clinic vs rheumatologist-led clinic

INTERVENTIONS:
Other: Nurse-led clinic vs rheumatologist-led clinic — The subjects are seeing a rheumatology nurse (experimental arm)instead of a rheumatologist (active comparator arm) after six months. Subjects in both arms are seeing a rheumatologist after 12 months and have the possibility to contact the rheumatology nurse.
  Other Names: Nurse-led clinic; Rheumatologist-led clinic

SUMMARY:
Randomized controlled trial including 100 subjects with rheumatic diseases and biological treatment with a 28 point-Disease Activity Score(DAS28)3.2 or less. The subjects will be randomized to either nurse-led clinic or rheumatologist-led clinic. The hypothesis is that there will be no difference in DAS28 between the two groups after 1 year follow-up.

DETAILED DESCRIPTION:
Aim To compare nurse-led clinic and rheumatologist-led clinic regarding results of treatment, and health economic costs.

Intervention Rheumatologist-led clinic: The subjects are seeing a rheumatologist after six months and after 12-months of intervention and have the possibility to contact the rheumatology clinic.

Nurse-led clinic: The subjects are seeing a rheumatology nurse after six months and a rheumatologist after 12 months of intervention and have the possibility to contact the rheumatology nurse during the intervention.

Outcome measures:

Main outcome: DAS28 and costs for the clinics respectively.

Secondary outcome: HAQ (Health Assessment Questionnaire), VAS-pain (Visual Analog Scale), VAS-global health, VAS-satisfaction, VAS-security/trust, Tender joints, swollen joints, Quality of life-EQ5D, Effective consumer survey 17, Inflammatory parameters in blood.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with rheumatologic diseases and biological treatment with a DAS28 of 3.2 or less

Exclusion Criteria:

* The subjects should not have problems with infections due to treatment
* Subjects with difficulties speaking and/or reading swedish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
DAS28 and costs for the clinics respectively. | Baseline at 0 months, 6 months, 12 months

SECONDARY OUTCOMES:
HAQ (Health Assessment Questionnaire), VAS-pain (Visual Analog Scale), VAS-global health, VAS-satisfaction, VAS-security/trust, Tender joints, swollen joints, Quality of life-EQ5D, Effective consumer survey 17, Inflammatory parameters in blood. | Baseline at 0 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Larsson, RN, PhD-stud, Principal Investigator — R&D-centre Spenshult; Stefan Bergman, MD, PhD, Study Director — R&D-centre Spenshult; Barbro Arvidsson, RNT, prof, Study Chair — R&D-centre Spenshult; Bengt Fridlund, RNT, prof, Study Chair — University of Jönköping, Sweden
Locations (1):
- Spenshult Hospital, Oskarström, Oskarström, Sweden

REFERENCES:
- [Derived] Larsson I, Fridlund B, Arvidsson B, Teleman A, Svedberg P, Bergman S. A nurse-led rheumatology clinic versus rheumatologist-led clinic in monitoring of patients with chronic inflammatory arthritis undergoing biological therapy: a cost comparison study in a randomised controlled trial. BMC Musculoskelet Disord. 2015 Nov 16;16:354. doi: 10.1186/s12891-015-0817-6. PMID 26573936
- See also: Related Info — http://www.fou-spenshult.se